CLINICAL TRIAL: NCT01769417
Title: A Phase 1, Randomized, Double-blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI4893, an Extended Half-Life Human Monoclonal Antibody Against Staphylococcus Aureus Alpha Toxin, in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI4893 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: CD-ID-MEDI4893-1133
Record Dates: First submitted 2013-01-11; First posted 2013-01-16 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections | interventions — suvratoxumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MEDI4893 (Active Comparator)
  Interventions: Drug: MEDI4893

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: MEDI4893 — Human immunoglobulin G1 kappa monoclonal antibody
  Other Names: Active comparator
  Arms: MEDI4893

SUMMARY:
This is a Phase 1, first time in human study enrolling approximately 33 healthy adult subjects (18-65 yrs) from one study site. The purpose of this study is to evaluate the safety, tolerability and PK of MEDI4893 in healthy adult volunteers administered as a single IV dose compared with placebo, across 4 cohorts. The 4 dose cohorts will enroll sequentially. Subjects will be followed for safety from the time of Informed Consent through 360 days post dose.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability and pharmacokinetics of MEDI4893, an extended half-life human monoclonal antibody against Staphylococcus aureus alpha toxin, in healthy adult subjects. Approximately 33 subjects will be enrolled across 4 fixed dose cohorts at 1 study site . This study will last approximately 389 days, constituting a screening period of up to 28 days, 1 day of investigational product administration, and a 360 day safety follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 65 years at screening.
2. Written informed consent and any locally required authorization (eg, HIPAA) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
3. Females of childbearing age using contraception for at least 28 days prior to receiving the dose of investigational product, and for 1 year after receiving IP.
4. Weight ≥ 45 kg and ≤ 110 kg at screening.
5. Healthy by medical history and physical examination at screening.
6. Systolic blood pressure (BP) < 140 mm Hg and diastolic BP < 90 mm Hg at screening.
7. Normal electrocardiogram (ECG) at screening.
8. Able to complete the 360-day postdose follow-up period as required by the protocol.

Exclusion Criteria:

1. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
2. Employees of the sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
3. Acute illness at study entry.
4. Fever 99.5F or higher on day of dosing.
5. Any drug therapy within 7 days prior to Day 1.
6. Blood donation in excess of 400 mL within 6 months prior to study entry.
7. Receipt of immunoglobulin or blood products within 6 months prior to study entry.
8. Receipt of any prior investigational drug or investigational vaccine within 120 days prior to investigational product dosing or planned dosing
9. Receipt of any standard vaccine within 14 days prior to investigational product dosing.
10. Previous receipt of a monoclonal antibody.
11. Receipt of immunosuppressive medications in the prior year or any active or prior history of immunodeficiency. Any course of systemic corticosteroids of more than 7 day duration during the prior year excludes a subject.
12. History of allergic disease or reactions likely to be exacerbated by any component of the investigational product.
13. Previous medical history or evidence of an intercurrent illness that may compromise the safety of the subject in the study.
14. Evidence of any systemic disease on physical examination at screening.
15. Evidence of infection (ie, positive laboratory test result) with hepatitis A, B, or C virus or human immunodeficiency virus (HIV) at screening.
16. Any of the following at screening:

    1. Hemoglobin < 12.0 g/dL for males and < 11.5 g/dL for females.
    2. WBC count < 3,800/mm3.
    3. Platelet count < 140,000/mm3.
    4. AST, ALT, BUN, serum creatinine > upper limit of normal (ULN).
    5. Positive Urine Class A drug screen.
    6. Other abnormal laboratory values in the screening panel, which in the opinion of the principal investigator, are judged to be clinically significant or potentially confound study results.
17. Pregnant or nursing mother.
18. Active alcohol or drug abuse or history of alcohol or drug abuse that, in the opinion of the principal investigator, might compromise subject safety, study safety assessments, or ability of subject to comply with study requirements.
19. Concurrent enrollment in another interventional study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The occurence of adverse events and serious adverse events. | From the time of informed consent through 360 days post dose
Vital Sign Measurements | Pre-dose through Study Day 15
  blood pressure, heart rate, respiratory rate, temperature
Clinical Safety lab measurements | from Day 1 (pre-dose) through 90 days post dose
  Chemistry, Hematology and urinalysis

SECONDARY OUTCOMES:
Pharmacokinetic Assessments - Serum | Pre-dose through 360 days post dose
  MEDI4893 Pharmacokinetic parameters.
Anti Drug Antibody (ADA) Assessments - Serum | Pre-dose through 360 days post dose
  ADA responses to MEDI4893.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Schwartz, M.D., Principal Investigator — Research Site; Hasan Jafri, M.D., Study Director — MedImmune LLC
Locations (1):
- Research Site, Miami, Florida, United States